CLINICAL TRIAL: NCT01051531
Title: Safety, Tolerability, and Treatment Response of Paliperidone Palmitate in Subjects With Schizophrenia When Switching From Oral Antipsychotics
Brief Title: A Safety, Tolerability, and Treatment Response Study of Paliperidone Palmitate Administered to Patients With Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR016522; R092670SCH3009 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2010-01-07; First posted 2010-01-18 (Estimated); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; R092670; Paliperidone palmitate; Diagnostic and Statistical Manual of Mental Disorders, 4th Edition; Intramuscular injection
MeSH Terms: conditions — Schizophrenia; Disease | interventions — Paliperidone Palmitate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

ARMS (1):
- Paliperidone palmitate (Experimental)
  Interventions: Drug: Paliperidone palmitate

INTERVENTIONS:
Drug: Paliperidone palmitate — One intramuscular (IM) injection of paliperidone palmitate 150 mg equivalent (eq.) on Day 1, 100 mg eq. on Day 8, and 75 mg eq. on Day 38. Thereafter, one IM injection of paliperidone palmitate 50, 75, 100, or 150 mg eq. once monthly. Doses may be adjusted every 30 days per the clinician's judgment within the dose range of 50 to 150 mg eq.

SUMMARY:
The purpose of the study is to evaluate the safety, tolerability and treatment response of paliperidone palmitate administered as once-monthly injections to patients with schizophrenia.

DETAILED DESCRIPTION:
This study is an 18-month, single-group, open-label (name of study drug is known to patients), multicenter study to evaluate the safety, tolerability and treatment response of paliperidone palmitate administered as once-monthly injections to patients with schizophrenia who previously received treatment with oral antipsychotic medications. A target of 587 patients (inpatients or outpatients) with schizophrenia will be enrolled in the study and will receive, without cost, injections of study drug (paliperidone palmitate) on Days 1, 8, 38, and thereafter at one-month intervals up to 18 months. Enrollment in the study will be limited to patients who are diagnosed with schizophrenia within the past 5 years. The study will consist of a screening period of up to 5 days before treatment, an 18-month treatment period, and an end-of-study or early withdrawal visit approximately 30 days after the last injection of study drug. During the screening period (after patients have provided signed informed consent to participate in the study), information will be collected regarding the patients medical and psychiatric history, demographics (age and race), current symptoms of the patients schizophrenia, and whether or not the patient would like to sign an additional informed consent form to participate in the pharmacogenomic (the study of how genes affect a person's response to drugs) component of the study that involves the collection of one 10 ml blood sample (equivalent to about 2 teaspoons of blood). During screening, entry criteria for the study will be reviewed and a physical examination performed. Patients will also be asked questions about the types of healthcare resources (institutionalizations/hospitalizations, emergency room visits, etc) they utilized during the previous 12 months however, this information is optional and its collection will depend upon the availability of the data. Patients who are currently receiving treatment with any oral antipsychotic medication must discontinue the use of the medication by Day 1 of the study. If the patient was receiving a high dose of an antipsychotic medication or was also receiving an anticholinergic medication (a drug that prevents involuntary muscle movements associated with the use of antipsychotic drugs in the treatment of schizophrenia), the investigator may decide to have the patients dose of antipsychotic (and/or anticholinergic) medication tapered (gradually reduced) to discontinuation beginning on Day 1. The patients time to taper-off the previous antipsychotic and/or anticholinergic medications will depend on the dose of the medication. Patients receiving anxiolytics (anti-anxiety drugs), mood stabilizers, anticholinergics, or antidepressants greater than 4 weeks before the screening visit will be allowed to continue taking these drugs. Upon meeting the entry criteria for the study, patients will receive a total of 19 intramuscular (IM) injections of paliperidone palmitate during the 18-month treatment period as follows: 150 mg equivalent (eq) on Day 1, 100 mg eq on Day 8, 75 mg eq on Day 38, and paliperidone palmitate injections of 50, 75, 100, or 150 mg eq once monthly on Days 68, 98, 128, 158, 188, 218, 248, 278, 308, 338, 368, 398, 428, 458, 488 and 518. Depending on the patients ability to tolerate a dose paliperidone palmitate, doses may be adjusted higher or lower every 30 days per the clinicians judgment within the dose range of 50 to 150 mg eq. If the patient reports any signs or symptoms of worsening of schizophrenia, the investigator may prescribe a rescue medication (quick-relief or fast-acting medications that usually work right away to relieve symptoms) such as lorazepam (an antianxiety drug) to control agitation, irritability, restlessness, and hostility. The investigator may also prescribe an anticholinergic medication to treat involuntary movement disorders if observed in patients. All prescription and over-the-counter medications taken by patients during the study are to be reported. At the end of the 18-month treatment period, all patients will complete an end-of-study visit (or early withdrawal visit for patients who do not complete the study) to have a physical examination performed, laboratory tests (including a urine pregnancy test for women of childbearing potential) performed, vital signs measured, and information collected regarding the occurrence of adverse events and the use of medications other than study drug from the time of the previous study visit to the end-of-study (or early withdrawal visit). The primary objective of the study is to evaluate safety, tolerability and treatment response of once-monthly injections of paliperidone palmitate measured by the use of a Positive And Negative Symptom Scale (PANSS). The safety and tolerability of once-monthly injections of paliperidone palmitate administered to patients with schizophrenia will be evaluated during the study by monitoring adverse events, findings from clinical laboratory tests (serum chemistry including lipids), vital sign measurements (blood pressure, pulse rate, and weight), physical examinations, and movement disorder evaluations using the Extrapyramidal Symptom Rating Scale [ESRS-A]). All clinically significant abnormalities in patients that persist at the end of the study will be followed by the Investigator until resolution or until a clinically stable endpoint is reached. Treatment response will be evaluated 5 times during the study (Visits 2, 4, 6, 8 and 10) by findings obtained from the PANSS (a 30-item questionnaire that is administered to the patient by a qualified person [ie, rater] to measure the presence/absence and severity of positive and negative symptoms of schizophrenia. In addition to the safety, tolerability, and treatment response data collected, patients who volunteer to participate in the pharmacogenomic component of the study will have one 10 ml sample of blood collected at on Days of Visit 2. If a replacement blood sample is needed for the pharmacogenomic component of the study, the patient will need to sign an additional informed consent form. Patients will receive a paliperidone palmitate intramuscular (IM) injection of 150 mg equivalent (eq) on Day 1, 100 mg eq on Day 8, and 75 mg eq on Day 38.Thereafter, patients will receive once monthly IM injections of 50, 75, 100, or 150 mg eq of paliperidone palmitate. Doses may be adjusted every 30 days per the clinician's judgment within the dose range of 50 to 150 mg eq.Patients will receive a total of 19 injections of study drug over an 18-month treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent to participate in the study obtained
* Signed informed consent to participate in the optional pharmacogenomic component of the study obtained (refusal to give consent for the pharmacogenomic component of the study does not exclude a patient from participation in the clinical study)
* Confirmation of diagnosis of schizophrenia according to the Diagnostic and Statistical Manual of Mental Disorders, 4th Edition (DSM-IV) within 5 years prior to screening
* Patient is willing and able to fill out self-administered questionnaires during the study
* confirmation that patient has been given an adequate dose of an appropriate oral antipsychotic for an adequate period of time before enrollment, but previous treatment is considered unsuccessful due to one or more of the following reasons: lack of efficacy, lack of tolerability or safety, lack of compliance and/or other reasons to switch to another antipsychotic medication

Exclusion Criteria:

* The patient's psychiatric diagnosis is due to the direct pharmacological effects of a drug of abuse substance or medication, or is due to a general medical condition (eg, clinically notable hypothyroidism)
* The patient is treatment resistant in the judgment of the investigator
* The patient meets the DSM-IV definition of substance dependence (except for nicotine and caffeine) within 6 months prior to entry
* The patient has a previously defined hypersensitivity (anaphylaxis-type reaction) to risperidone or paliperidone or excipients
* The patient has received treatment with a long-acting injectable antipsychotic within 3 injection cycles prior to baseline, received clozapine within 3 months prior to screening, received treatment with other investigational agents within 30 days of the screening visit, has participated in more than one investigational drug study in the past 12 months, or has planned use of other investigational drugs during the time frame of the study
* History or current symptoms of tardive dyskinesia, history of neuroleptic malignant syndrome, or evidence of clinically significant cardiovascular, renal, hepatic, gastrointestinal, neurological, endocrine, metabolic or pulmonary disease in the past 6 months

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 546 (Actual)
Dates: Start 2010-04-22 (Actual); Primary Completion 2013-05-17 (Actual); Study Completion 2013-05-17 (Actual)

PRIMARY OUTCOMES:
Treatment response will be evaluated by findings from the PANSS-a 30-item questionnaire that is administered to the patient by a qualified person (ie, rater) to measure the presence/absence and severity of positive and negative symptoms of schizophrenia | Treatment response will be evaluated at 5 times during the study (Day 1, day 38, day 98, day 188, day 368 and day 548).

SECONDARY OUTCOMES:
The change in personal and social performance (PSP) score and evolution of ratio of mild degree dysfunction, varying degree difficulty, and poor level function based on PSP score after switch to paliperidone palmitate | 5 visits (Day 1, day 38, day 188, day 368 and day 548)
The rate of discontinuation, the rate of patients hospitalized, the total number and mean duration of institutionalizations, the overall score in global severity of illness, symptom remission, and medication satisfaction questionnaire findings | 9 visits (Day 1, day 8, day 38, day 98, day 188, day 278, day 368, day458 and day 548)
The changes in total PANSS score and PANSS sub-domains/symptom factors | 5 visits (Day 1, day 38, day 188, day 368 and day 548).
Safety measures (laboratories, adverse events, ESRS-A) | Laboratories (Days 1 and 548; Adverse events (Days 1, 8,38,68,98,128,158,188,218,248, 278, 308, 338, 368, 398, 448, 458, 488, 518 and 548) ESRS-A (Days 1, 8, 38, 98, 188, 278, 368, 458 and 548)
Assessment of healthcare resource utilization | 7 visits (Day -7, Day 98, day 188, day 278, day 368, day 458 and day 548)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (41):
- Australia (9):
  - Dandenong
  - Elizabeth Vale
  - Epping
  - Frankston
  - Glenside
  - Heidelberg
  - Melbourne
  - Prahran
  - Westmead
- China (5):
  - Beijing
  - Guangzhou
  - Nanjing
  - Shanghai
  - Xi'an
- Hong Kong, Hong Kong
- Malaysia (7):
  - Johor Bahru
  - Kota Bharu
  - Kota Kinabalu
  - Kuala Lumpur
  - Kuching
  - Tanjong Rambutan
  - Terengganu
- Auckland, New Zealand
- Philippines (2):
  - Pasig
  - Pasig National Capitol Region
- South Korea (7):
  - Busan
  - Daegu
  - Daejeon
  - Gwangju
  - Gyeonggi-do
  - Incheon
  - Seoul
- Taiwan (5):
  - Changhua County
  - Kaohsiung City
  - Taichung
  - Tainan
  - Taipei
- Thailand (4):
  - Bangkok
  - Khon Kaen
  - Songkhla
  - Ubon Ratchathani

REFERENCES:
- See also: Safety, Tolerability, and Treatment Response of Paliperidone Palmitate in Subjects with Schizophrenia When Switching from Oral Antipsychotics — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=691&filename=CR016522_CSR.pdf